CLINICAL TRIAL: NCT04580303
Title: A Phase 2 Multicenter, Open-label, Randomized, Parallel-group, Multiple-dose Study to Assess the Effectiveness, Safety and Satisfaction With Collagenase Clostridium Histolyticum Grid Technique Injections of Buttock or Thigh Cellulite With Laxity in Adult Females
Brief Title: CCH Treatment of Cellulite in the Presence of Dermal Laxity With Comparison Between Two (2) Different Injection Techniques
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN3835-224
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-08

CONDITIONS: Edematous Fibrosclerotic Panniculopathy; Cellulite; Laxity; Skin
MeSH Terms: conditions — Cellulite; Cutis Laxa | interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Uniform 0.1-milliliters (mL) 1-Aliquot Grid Injection Technique (Buttock) (Active Comparator): Dose per participant per treatment visit = up to 1.68 milligrams (mg) of CCH (0.84 mg in each treatment area)
  Interventions: Drug: collagenase clostridium histolyticum
- Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttock) (Active Comparator): Dose per participant per treatment visit = up to 1.68 mg of CCH (0.84 mg in each treatment area)
  Interventions: Drug: collagenase clostridium histolyticum
- Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Thigh) (Active Comparator): Dose per participant per treatment visit = up to 1.68 mg of CCH (0.84 mg in each treatment area)
  Interventions: Drug: collagenase clostridium histolyticum
- Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Thigh) (Active Comparator): Dose per participant per treatment visit = up to 1.68 mg of CCH (0.84 mg in each treatment area)
  Interventions: Drug: collagenase clostridium histolyticum

INTERVENTIONS:
Drug: collagenase clostridium histolyticum — Delivered via uniform grid injection techniques.
  Other Names: EN3835; CCH

SUMMARY:
This study is designed to investigate the safety and efficacy of collagenase clostridium histolyticum (CCH) for the treatment of mild to moderate edematous fibrosclerotic panniculopathy (cellulite) in participants with moderate to severe dermal laxity in the buttocks or thighs with comparison between two (2) different CCH injection techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Have a body mass index of 18 to <29.9 kilograms/square meters
2. Have either both buttocks or both posterolateral thighs with:

   1. Score of 2 or 3 (mild or moderate cellulite) as reported by the investigator using the Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS)
   2. Hexsel Cellulite Severity Scale (CSS) Subsection D "Grade of Laxity, Flaccidity, or Sagging Skin" score of 2 or 3 (moderate or severe) as determined by the investigator
3. Have a negative pregnancy test or be of non-childbearing potential
4. Be willing and able to cooperate with the requirements of the study
5. Be willing to apply sunscreen to the treatment areas before each exposure to the sun for the duration of the study (from the Screening Visit through the Day 180/Early Termination Visit).

Exclusion Criteria:

1. Has a history of hypersensitivity or allergy to collagenase or any other excipients of CCH.
2. During Screening has a CR-PCSS score of less than 2 or greater than 3 for the area to be treated (buttocks or thighs) and/or has a Hexsel CSS Subsection D "Grade of Laxity, Flaccidity, or Sagging Skin" score of less than 2 or greater than 3 (severe) for the areas to be treated (buttocks or thighs).
3. Has a coagulation disorder, which requires anticoagulant or antiplatelet medication during the study (except for ≤150 mg aspirin daily), or has taken anticoagulant or antiplatelet medication(s) within 14 days before injection of study treatment (except for ≤150 mg aspirin daily).
4. Is a prisoner, an individual with impaired decision making capacity, employees (temporary, part-time, full-time, etc) or a family member of the research staff conducting the study, or of the sponsor, or of the contract research organization, or of the Institutional Review Board (IRB)/Independent Ethics Committee (IEC), or in the judgment of the investigator the participant is disadvantaged and vulnerable to coercion due to lack of education, or due to poor economic circumstances.
5. Has received any collagenase treatments at any time prior to treatment in this study and/or has received EN3835 or CCH in a previous investigational study for cellulite.
6. Is pregnant and/or is breast-feeding or plans to become pregnant and/or to breast-feed during the course of the study.
7. Has a history of scarring due to keloids or abnormal wound healing.
8. Has local (in areas to be treated) conditions (thrombosis, vascular disorder, active infection/inflammation, active cutaneous alteration, tattoo/mole) that restricts study participation
9. Has history of drug or alcohol abuse within the 5 years prior to the Screening Visit.
10. Has evidence of clinically significant abnormalities, as judged by the investigator, in any of the following: physical examination findings, electrocardiogram (ECG), clinical laboratory values, or vital signs.

    The sponsor's medical monitor will be required to review the results for confirmation of eligibility in the case of any of the following: abnormalities in electrocardiograms indicating corrected QT interval (QTc) prolongation of 470 milliseconds or greater; and clinical laboratory values of liver enzymes
11. Has used or intends to use any of the local application/therapies/injections/procedures that restricts study participation.
12. Has any other condition(s) that, in the investigator's opinion, might indicate the participant to be unsuitable for the study.
13. For the subset of participants participating in the collection of ultrasound data, the following exclusions will apply: participants will be excluded who have: a history of a spinal laminectomy, a previous history or presence of vascular abnormalities (for example, deep vein thrombosis, thrombophlebitis), a healing fracture, an impaired sensation within, or near, the planned treatment area, or any implants within, or near, the planned treatment area.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 35 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hernandez, Study Director — Endo Pharmaceuticals
Locations (3):
- United States (3):
  - Endo Clinical Trial Site #3, Coral Gables, Florida
  - Endo Clinical Trial Site #2, Metairie, Louisiana
  - Endo Clinical Trial Site #1, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive treatment in either a uniform 0.1-milliliter (mL), 1-aliquot, grid injection technique or uniform 0.3-mL, 2-aliquot grid injection technique in a 1:1 ratio. Each participant had 2 treatment areas (each buttock or each thigh).
Units Other Than Participants: buttock or thigh
Groups:
- Uniform 0.1-mL (Milliliter) 1-Aliquot Grid Injection Technique (Buttocks): Dose per participant per treatment visit = up to 1.68 milligrams (mg) of collagenase clostridium histolyticum (CCH) (0.84 mg in each treatment area).
- Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttocks); Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Thighs); Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Thighs): Dose per participant per treatment visit = up to 1.68 mg of CCH (0.84 mg in each treatment area).
Period: Overall Study
Arm/Group | Uniform 0.1-mL (Milliliter) 1-Aliquot Grid Injection Technique (Buttocks) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttocks) | Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Thighs) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Thighs)
Started | 7; 14 buttock or thigh | 9; 18 buttock or thigh | 9; 18 buttock or thigh | 10; 20 buttock or thigh
Completed | 7; 14 buttock or thigh | 8; 16 buttock or thigh | 8; 16 buttock or thigh | 10; 20 buttock or thigh
Not Completed | 0; 0 buttock or thigh | 1; 2 buttock or thigh | 1; 2 buttock or thigh | 0; 0 buttock or thigh
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All enrolled participants who received at least 1 injection of CCH. Participants who received injection in the buttock or thigh are combined for each injection technique.
Groups:
- Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Buttock or Thigh); Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttock or Thigh): Dose per participant per treatment visit = up to 1.68 mg of CCH (0.84 mg in each treatment area).
- Total: Total of all reporting groups
Arm/Group | Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Buttock or Thigh) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttock or Thigh) | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.73 (8.844) | 42.51 (6.225) | 41.70 (7.472)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 13 | 18 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of 1-Level Responders (+1 or Better Score) on the Investigator-Global Aesthetic Improvement Scale (I-GAIS) for Either Buttock or Either Thigh
Description: I-GAIS is a 7-point scale rating global aesthetic improvement in appearance, compared to pretreatment, as judged by the investigator ranging from "Very Much Worse" (-3), "Much Worse" (-2), "Worse" (-1), "No Change" (0), "Improved" (+1), "Much Improved" (+2), and "Very Much Improved" (+3). One-level I-GAIS Responder for a treatment area (left buttock, right buttock, left thigh, or right thigh) was defined as any participant with an improved (+1, +2 or +3) score on the I-GAIS at the analysis visit for that treatment area. The percentage of participants who were 1-level responders for either buttock (right or left) or either thigh (right or left) is presented.
Time Frame: Day 180
Population: Modified Intent-to-Treat (mITT) Population: All enrolled participants who received at least 1 injection of CCH and who had at least 1 valid I-GAIS evaluation after the injection of CCH.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Buttocks); Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttocks); Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Thighs); Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Thighs): Dose per participant per treatment visit = up to 1.68 mg of CCH (0.84 mg in each treatment area).
Arm/Group | Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Buttocks) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttocks) | Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Thighs) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Thighs)
Number analyzed (Participants) | 7 | 8 | 8 | 10
percentage of participants | 85.7 [42.13 to 99.64] | 87.5 [47.35 to 99.68] | 75.0 [34.91 to 96.81] | 80.0 [44.39 to 97.48]

2. Secondary Outcome: Percentage of 1-Level Responders (+1 or Better Score) on the I-GAIS for Either Buttock or Either Thigh
Description: as for outcome 1
Time Frame: Days 28, 56, 84, 112, and 140
Population: mITT Population: All enrolled participants who received at least 1 injection of CCH and who had at least 1 valid I-GAIS evaluation after the injection of CCH.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Buttocks) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttocks) | Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Thighs) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Thighs)
Number analyzed (Participants) | 7 | 9 | 9 | 10
percentage of participants
  Day 28: number analyzed (Participants) | 7 | 9 | 9 | 9
  Day 28 | 71.4 [29.04 to 96.33] | 44.4 [13.70 to 78.80] | 77.8 [39.99 to 97.19] | 77.8 [39.99 to 97.19]
  Day 56: number analyzed (Participants) | 7 | 8 | 9 | 9
  Day 56 | 85.7 [42.13 to 99.64] | 62.5 [24.49 to 91.48] | 88.9 [51.75 to 99.72] | 88.9 [51.75 to 99.72]
  Day 84: number analyzed (Participants) | 7 | 8 | 9 | 10
  Day 84 | 57.1 [18.41 to 90.10] | 75.0 [34.91 to 96.81] | 77.8 [39.99 to 97.19] | 70.0 [34.75 to 93.33]
  Day 112: number analyzed (Participants) | 7 | 8 | 9 | 10
  Day 112 | 85.7 [42.13 to 99.64] | 50.0 [15.70 to 84.30] | 77.8 [39.99 to 97.19] | 80.0 [44.39 to 97.48]
  Day 140: number analyzed (Participants) | 7 | 8 | 8 | 10
  Day 140 | 71.4 [29.04 to 96.33] | 75.0 [34.91 to 96.81] | 75.0 [34.91 to 96.81] | 80.0 [44.39 to 97.48]

3. Secondary Outcome: Percentage of 1-Level Responders (+1 or Better Score) on the Subject Global Aesthetic Improvement Scale (S-GAIS) for Either Buttock or Either Thigh
Description: S-GAIS assessments were based on digital photographs, and were performed separately for each of 2 treatment areas. S-GAIS is a 7-point scale rating global aesthetic improvement in appearance, compared to pretreatment, as judged by the participant ranging from "Very Much Worse" (-3), "Much Worse" (-2), "Worse" (-1), "No Change" (0), "Improved" (+1), "Much Improved" (+2), and "Very Much Improved" (+3). One-level S-GAIS Responder for a treatment area (left buttock, right buttock, left thigh, or right thigh) was defined as any participant with an improved (+1, +2 or +3) score on the S-GAIS at the analysis visit for that treatment area. The percentage of participants who were 1-level responders for either buttock (right or left) or either thigh (right or left) is presented.
Time Frame: Days 28, 56, 84, 112, 140, and 180
Population: mITT Population: All enrolled participants who received at least 1 injection of CCH and who had at least 1 valid S-GAIS evaluation after the injection of CCH.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Buttocks) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttocks) | Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Thighs) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Thighs)
Number analyzed (Participants) | 7 | 9 | 9 | 10
percentage of participants
  Day 28: number analyzed (Participants) | 7 | 9 | 9 | 9
  Day 28 | 71.4 [29.04 to 96.33] | 44.4 [13.70 to 78.80] | 66.7 [29.93 to 92.51] | 66.7 [29.93 to 92.51]
  Day 56: number analyzed (Participants) | 7 | 8 | 9 | 9
  Day 56 | 85.7 [42.13 to 99.64] | 75.0 [34.91 to 96.81] | 88.9 [51.75 to 99.72] | 88.9 [51.75 to 99.72]
  Day 84: number analyzed (Participants) | 7 | 8 | 9 | 10
  Day 84 | 71.4 [29.04 to 96.33] | 87.5 [47.35 to 99.68] | 55.6 [21.20 to 86.30] | 70.0 [34.75 to 93.33]
  Day 112: number analyzed (Participants) | 7 | 8 | 9 | 10
  Day 112 | 85.7 [42.13 to 99.64] | 62.5 [24.49 to 91.48] | 55.6 [21.20 to 86.30] | 70.0 [34.75 to 93.33]
  Day 140: number analyzed (Participants) | 7 | 8 | 8 | 10
  Day 140 | 71.4 [29.04 to 96.33] | 87.5 [47.35 to 99.68] | 62.5 [24.49 to 91.48] | 70.0 [34.75 to 93.33]
  Day 180: number analyzed (Participants) | 7 | 8 | 8 | 10
  Day 180 | 85.7 [42.13 to 99.64] | 100.0 [NA to NA] — Confidence interval was not calculated for dispersion since all participants were responders. | 62.5 [24.49 to 91.48] | 90.0 [55.50 to 99.75]

4. Secondary Outcome: Change From Baseline in Body-Q Appraisal of Cellulite Total Score
Description: The Body-Q Appraisal of Cellulite is a subset of 11 questions from the Body-Q questionnaire developed to measure participant perceptions of weight loss and/or body contouring. Total score is the sum of all 11 question scores. The minimum possible total score is 11 and the maximum possible total score is 44. Higher scores indicate the individual is less bothered by their cellulite.
Time Frame: Baseline, Day 180
Population: mITT Population: All enrolled participants who received at least 1 injection of CCH and who had an assessment as the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Buttocks) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttocks) | Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Thighs) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Thighs)
Number analyzed (Participants) | 7 | 8 | 8 | 10
units on a scale | 13.4 (11.12) | 13.6 (9.94) | 10.0 (5.81) | 6.4 (10.56)

5. Secondary Outcome: Change From Baseline in Hexsel Cellulite Severity Scale (CSS) Subsection D Severity Score
Description: Hexsel CSS is a photonumeric scale that looks at 5 key morphologic features of cellulite using a 4-point scale from a low of 0 to high of 3: 0 (absence of laxity, flaccidity, or sagging skin), 1 (slight draped appearance), 2 (moderate draped appearance), and 3 (severe draped appearance). The investigator or qualified designee used the Hexsel CSS Subsection D to assess the severity of dermal laxity in each buttock or each thigh independently. A decrease from baseline indicated a better outcome.
Time Frame: Baseline, Days 28, 56, 84, 112,140, and 180
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Uniform 0.1-mL 1-Aliqout Grid Injection Technique (Buttocks); Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttocks); Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Thighs); Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Thighs): Dose per participant per treatment visit = up to 1.68 mg of CCH (0.84 mg in each treatment area).
Arm/Group | Uniform 0.1-mL 1-Aliqout Grid Injection Technique (Buttocks) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttocks) | Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Thighs) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Thighs)
Number analyzed (Participants) | 7 | 9 | 9 | 10
units on a scale
  Day 28 Left Treatment Area: number analyzed (Participants) | 6 | 9 | 9 | 9
  Day 28 Left Treatment Area | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Day 28 Right Treatment Area: number analyzed (Participants) | 6 | 9 | 9 | 9
  Day 28 Right Treatment Area | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Day 56 Left Treatment Area: number analyzed (Participants) | 7 | 8 | 9 | 9
  Day 56 Left Treatment Area | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Day 56 Right Treatment Area: number analyzed (Participants) | 7 | 8 | 9 | 9
  Day 56 Right Treatment Area | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Day 84 Left Treatment Area: number analyzed (Participants) | 7 | 8 | 9 | 10
  Day 84 Left Treatment Area | -0.1 (0.38) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Day 84 Right Treatment Area: number analyzed (Participants) | 7 | 8 | 9 | 10
  Day 84 Right Treatment Area | -0.1 (0.38) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Day 112 Left Treatment Area: number analyzed (Participants) | 7 | 8 | 9 | 10
  Day 112 Left Treatment Area | -0.1 (0.38) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Day 112 Right Treatment Area: number analyzed (Participants) | 7 | 8 | 9 | 10
  Day 112 Right Treatment Area | -0.1 (0.38) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Day 140 Left Treatment Area: number analyzed (Participants) | 7 | 8 | 8 | 10
  Day 140 Left Treatment Area | -0.4 (0.53) | -0.1 (0.35) | 0.0 (0.00) | -0.2 (0.42)
  Day 140 Right Treatment Area: number analyzed (Participants) | 7 | 8 | 8 | 10
  Day 140 Right Treatment Area | -0.3 (0.49) | -0.1 (0.35) | -0.1 (0.35) | -0.2 (0.42)
  Day 180 Left Treatment Area: number analyzed (Participants) | 7 | 8 | 8 | 10
  Day 180 Left Treatment Area | -0.3 (0.49) | -0.1 (0.64) | -0.1 (0.35) | -0.6 (0.52)
  Day 180 Right Treatment Area: number analyzed (Participants) | 7 | 8 | 8 | 10
  Day 180 Right Treatment Area | -0.3 (0.49) | -0.1 (0.64) | -0.1 (0.35) | -0.5 (0.53)

6. Secondary Outcome: Percentage of Participants Positive for Anti-AUX-I and Anti-AUX-II Antibodies
Description: Blood samples were collected to assess anti-clostridial class I collagenase (AUX-I) and anti-Clostridial class II collagenase (AUX-II) antibody levels. The percentage of participants who were positive for anti-AUX-I and anti-AUX-II antibodies are presented.
Time Frame: Day 180
Population: mITT Population: All enrolled participants who received at least 1 injection of CCH and were assessed for anti-AUX-I and anti-AUX-II Antibodies at the specified timepoint. Immunogenicity analysis was conducted by overall participants and not treatment area/injection technique.
Measure: Number; unit: percentage of participants
Groups:
- CCH: Overall Participants: Participants who received CCH by either injection technique (1 aliquot or 2 aliquot grid techniques) in the buttocks or thighs.
Arm/Group | CCH: Overall Participants
Number analyzed (Participants) | 32
percentage of participants
  Anti-AUX-I Antibodies | 100
  Anti-AUX-II Antibodies | 100

7. Secondary Outcome: Percentage of Participants Positive for Neutralizing Antibodies to AUX-I and AUX-II
Description: Blood samples were collected to assess neutralizing antibodies to AUX-I and AUX-II. The percentage of participants who were positive for neutralizing antibodies to AUX-I and AUX-II are presented.
Time Frame: Day 180
Population: mITT Population: All enrolled participants who received at least 1 injection of CCH and who had an assessment as the specified timepoint. Immunogenicity analysis was conducted by overall participants and not treatment area/injection technique.
Measure: Number; unit: percentage of participants
Arm/Group | CCH: Overall Participants
Number analyzed (Participants) | 32
percentage of participants
  Neutralizing antibodies to AUX-I | 87.5
  Neutralizing antibodies to AUX-II | 84.4

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through Day 180
Description: Safety Population: All enrolled participants who received at least 1 injection of CCH. Adverse events are reported by participant and not treatment area. Participants who received injection in the either the buttocks or thighs are combined for each injection technique.
Groups:
- Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Buttocks or Thighs); Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttocks or Thighs): Dose per participant per treatment visit = up to 1.68 mg of CCH (0.84 mg in each treatment area).
Arm/Group | Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Buttocks or Thighs) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttocks or Thighs)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19
Other Adverse Events (participants affected / at risk) | 16/16 | 19/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Uniform 0.1-mL 1-Aliquot Grid Injection Technique (Buttocks or Thighs) (N=16) | Uniform 0.3-mL 2-Aliquot Grid Injection Technique (Buttocks or Thighs) (N=19)
Fatigue (General disorders) | 0 | 1
Implant site inflammation (General disorders) | 0 | 1
Implant site pain (General disorders) | 0 | 1
Injection site bruising (General disorders) | 16 | 19
Injection site discolouration (General disorders) | 1 | 1
Injection site mass (General disorders) | 0 | 1
Injection site pain (General disorders) | 10 | 13
Injection site pruritus (General disorders) | 2 | 2
Injection site swelling (General disorders) | 10 | 10
Injection site urticaria (General disorders) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Device breakage (Product Issues) | 0 | 1
Alcoholism (Psychiatric disorders) | 1 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT04580303/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT04580303/SAP_001.pdf